CLINICAL TRIAL: NCT05988606
Title: Acute Work Rate Adjustments During High-intensity Interval Training in a Hot and Temperate Environment
Brief Title: Work Rate Adjustments During a High-intensity Interval Training on a Stationary Bike in a Hot and Temperate Environment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 21-02-4359
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: High-Intensity Interval Training; Heat
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Participants completed all trials and were compared to themselves.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 15TEMP (Experimental): Participants cycled at 70% heart rate max for 8 min as a warm-up and then completed one round of HIIT, i.e., 4 min at 90% heart rate max followed by 3 min at 70% heart rate max for a total of 15 minutes in a temperate environment, followed by a graded exercise test to measure maximal aerobic capacity.
  Interventions: Behavioral: 15 minutes of high-intensity interval training; Other: Temperate environment
- 15HEAT (Experimental): Participants cycled at 70% heart rate max for 8 min as a warm-up and then completed one round of HIIT, i.e., 4 min at 90% heart rate max followed by 3 min at 70% heart rate max for a total of 15 minutes in a hot environment, followed by a graded exercise test to measure maximal aerobic capacity.
  Interventions: Behavioral: 15 minutes of high-intensity interval training; Other: Hot environment
- 43TEMP (Experimental): Participants cycled at 70% heart rate max for 8 min as a warm-up and then performed the HIIT protocol (4 min at 90% heart rate max and 3 min at 70% heart rate max, repeated 4 times for a total of 43 minutes) in a temperate environment followed by a graded exercise test to measure maximal aerobic capacity.
  Interventions: Behavioral: 43 minutes of high-intensity interval training; Other: Temperate environment
- 43HEAT (Experimental): Participants cycled at 70% heart rate max for 8 min as a warm-up and then performed the HIIT protocol (4 min at 90% heart rate max and 3 min at 70% heart rate max, repeated 4 times for a total of 43 minutes) in a hot environment followed by a graded exercise test to measure maximal aerobic capacity.
  Interventions: Behavioral: 43 minutes of high-intensity interval training; Other: Hot environment
- Control (No Intervention): Participants completed a graded exercise test on a stationary bicycle in a temperate environment (~ 22 °C (72 °F), ~40% RH) to measure maximal aerobic capacity and maximal heart rate.

INTERVENTIONS:
Behavioral: 15 minutes of high-intensity interval training — Participants completed an 8 min warm-up and 1 round of high-intensity interval training
  Arms: 15HEAT; 15TEMP
Behavioral: 43 minutes of high-intensity interval training — Participants completed an 8 min warm-up and 5 rounds of high-intensity interval training
  Arms: 43HEAT; 43TEMP
Other: Hot environment — Participants exercised in a hot environment, ~ 35 °C, ~40% relative humidity.
  Arms: 15HEAT; 43HEAT
Other: Temperate environment — Participants exercised in a temperate environment, ~ 22 °C, ~40% relative humidity.
  Arms: 15TEMP; 43TEMP

SUMMARY:
The goal of this repeated measures study is to evaluate acute work rate adjustments during high-intensity interval training (HIIT) in a hot and temperate environment in healthy and active adults when using target heart rate to prescribe the exercise intensity.

The main questions it aims to answer are:

* Will HIIT based on target heart rate in a hot environment result in increased cardiovascular (i.e., elevated recovery HR) and thermal strain compared to HIIT in a temperate environment?
* Will work rate be lowered to a greater extent during HIIT in a hot environment compared to a temperate environment in order to maintain target heart rate?
* Will maximal aerobic capacity (V̇O2max) decrease to a greater extent after HIIT in the heat compared to a temperate environment?

Procedures:

Participants will complete 5 trials on a cycle ergometer. Trial 1 (Control Visit): Participants (n = 7) will have their maximal heart rate and V̇O2max measured in a temperate environment (~22 °C, 40% RH).

Experimental Trials 2-5: The order of the trials will be counterbalanced and randomly assigned to participants.

* 15TEMP: Participants will cycle at 70% of their maximum heart rate for 8 minutes as a warm-up, followed by one round of HIIT. The HIIT protocol consists of 4 minutes at 90% of maximum heart rate followed by 3 minutes at 70% of maximum heart rate, totaling 15 minutes, in a temperate environment (~22 °C, 40% RH). After the HIIT session, a graded exercise test will measure V̇O2max.
* 15HEAT: Similar to 15TEMP, but participants will perform the HIIT protocol in a hot environment (~35 °C, 40% RH).
* 43TEMP: Participants will cycle at 70% of their maximum heart rate for 8 minutes as a warm-up, followed by the HIIT protocol repeated four times (4 minutes at 90% of maximum heart rate and 3 minutes at 70% of maximum heart rate), totaling 43 minutes, in a temperate environment (~22 °C, 40% RH).
* 43HEAT: Similar to 43TEMP, but participants will perform the HIIT protocol in a hot environment (~35 °C, 40% RH).

ELIGIBILITY:
Inclusion Criteria:

* Participants were healthy males and females who are 18 to 39 years of age, recreationally active as defined by the American College of Sports Medicine, performing moderate-intensity aerobic exercise 30 min or more per session for at least 3 sessions per week for at least the past 3 months, and free of metabolic, cardiovascular, and renal disease

Exclusion Criteria:

* Individuals classified as needing medical clearance according to American College of Sports Medicine (ACSM) Guidelines were not allowed to participate. Needing medical clearance is defined by ACSM as 1) not being physically active and having known cardiovascular, metabolic, or renal disease and asymptomatic; 2) not being physically active and having any signs or symptoms suggestive of cardiovascular, metabolic, or renal disease; 3) participating in regular exercise and having known cardiovascular, metabolic, or renal disease and asymptomatic; or 4) participating in regular exercise and having any signs or symptoms suggestive of cardiovascular, metabolic, or renal disease .

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
Work rate adjustments | From the first work interval (min 9-12) to the last work interval (min 37-40).
  In a hot and temperate environment by how much does work rate need to be adjusted to maintain target heart rate?

SECONDARY OUTCOMES:
Cardiovascular strain | From the first recovery interval (min 13-15) to the last recovery interval (min 41-43).
  In a hot and temperate environment by how much does heart rate in the recovery intervals increase?
Thermal Strain | From the first work interval (min 9-12) to the last work interval (min 37-40).
  In a hot and temperate environment by how much do rectal temperature and skin temperature increase?
Maximal aerobic capacity | The end of the 15 min trials compared to the end of the 43 min trials.
  In a hot and temperate environment by how much does maximal aerobic capacity decrease?

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Alabama, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No